CLINICAL TRIAL: NCT00279812
Title: Selenium and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Food Standards Agency, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IFR02/2005; FSA 51949F (Other: Food Standards Agency)
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Immune response; Selenomethionine; Selenium enriched foods; Selenium status; Selenium biomarkers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 50ug selenium enriched yeast (Experimental): 50ug/d selenium enriched yeast (containing 60% selenomethionine)
  Interventions: Dietary Supplement: 50ug selenium enriched yeast
- 100ug selenium enriched yeast (Experimental): 100ug/d selenium enriched yeast (containing 60% selenomethionine)
  Interventions: Dietary Supplement: 100ug selenium enriched yeast
- 200ug selenium enriched yeast (Experimental): 200ug/d selenium enriched yeast (containing 60% selenomethionine)
  Interventions: Dietary Supplement: 200ug selenium enriched yeast
- Control onion (Experimental): 3 meals/wk containing un-enriched onions equivalent to 4ug/d Se
  Interventions: Dietary Supplement: Control onion
- Enriched onion (Experimental): 3 meals/wk containing enriched onions equivalent to 50ug/d Se
  Interventions: Dietary Supplement: Enriched onion

INTERVENTIONS:
Dietary Supplement: 50ug selenium enriched yeast — Selenomethionine supplement (50ug/d Se) for 12 weeks
  Arms: 50ug selenium enriched yeast
Dietary Supplement: 100ug selenium enriched yeast — Selenomethionine supplement (100ug/d Se) for 12 weeks
  Arms: 100ug selenium enriched yeast
Dietary Supplement: 200ug selenium enriched yeast — Selenomethionine supplement (200ug/d Se) for 12 weeks
  Arms: 200ug selenium enriched yeast
Dietary Supplement: Control onion — 3 meals per week containing un-enriched onion (4ug/d) for 12 weeks
  Arms: Control onion
Dietary Supplement: Enriched onion — 3 meals per week containing un-enriched onion (50ug/d) for 12 weeks
  Arms: Enriched onion
Other: Placebo — Placebo supplement for 12 weeks
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the relationship between dose and form of selenium on immune function, and to identify functional markers of selenium status.

DETAILED DESCRIPTION:
One of the proposed consequences of marginal selenium status is impaired immune function. Establishing the potential role of selenium as an enhancer of immune response in vivo may provide evidence-base for public health policy, with important consequences for preventing influenza and similar diseases in the elderly.

The project consists of a placebo controlled selenium supplementation study and a dietary intervention with un-enriched and selenium enriched onions. In a parallel group design, subjects will be given either one of three doses of Selenomethionine (50, 100 or 200µg selenium/day) or a placebo per day or selenium enriched or un-enriched onions (in the form of test meals) for 12 weeks. Changes in the expression of Se-responsive genes and proteins in blood will be measured and compared with changes in plasma Se concentration and selected selenoproteins. The relationship between dietary Se intake and systemic and mucosal immune responses to influenza vaccine will be examined. Changes in immune cell populations and the influence of Se on NK and CD8 cytotoxicity will be determined by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 50-64
* Plasma selenium level <1.2µmol/l (±10%)

Exclusion Criteria:

* Elevated blood pressure measurements (<90/50 or <95/50 if symptomatic or >160/100)
* Body mass index (BMI) <18.5 or >35
* Results of the clinical screening which are judged by the Human Nutrition Unit (HNU) Medical advisor to be indicative of a health problem and could compromise the well-being of the volunteer if they participated, or which would affect the data.
* Smokers
* Diagnosed with gastrointestinal disease (excluding hiatus hernia unless symptomatic or study intervention/procedure is contraindicated) for which they have been taking prescription drugs on a chronic basis.
* Diagnosed with a long-term illness requiring active treatment, e.g. diabetes, cancer, cardiovascular disease.
* On regularly prescribed medication known to have a profound effect on the immune function
* Regularly using antacids and laxatives (at least once a week)
* Sufferers of hay-fever taking regular steroid medication
* Unwillingness to discontinue dietary (other than vitamins and minerals) or herbal supplements less than one month prior to the start of the study and for the duration of the study
* Blood donation within 16 weeks of the first study sample and who intend to donate blood less than 16 weeks after the last study sample
* Antibiotic use within four weeks prior to starting the study
* Those who receive or plan to receive any other type of immunisation during the study period
* Those who have received an immunisation within 6 months of the start of the study
* Intention to go on holiday/trips for more than 2 weeks during the twelve week intervention
* Those planning a holiday/trip that requires immunisation during the twelve week intervention period
* Parallel participation in another research project which involves dietary intervention or sampling of biological fluids/materials
* Allergic to eggs or egg products
* Allergic to chicken protein
* Allergic to the antibiotic Gentamicin
* A history of Guillain-Barre syndrome

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2005-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Fairweather-Tait, PhD, Principal Investigator — University of East Anglia
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Ivory K, Prieto E, Spinks C, Armah CN, Goldson AJ, Dainty JR, Nicoletti C. Selenium supplementation has beneficial and detrimental effects on immunity to influenza vaccine in older adults. Clin Nutr. 2017 Apr;36(2):407-415. doi: 10.1016/j.clnu.2015.12.003. Epub 2015 Dec 24. PMID 26803169
- [Derived] Goldson AJ, Fairweather-Tait SJ, Armah CN, Bao Y, Broadley MR, Dainty JR, Furniss C, Hart DJ, Teucher B, Hurst R. Effects of selenium supplementation on selenoprotein gene expression and response to influenza vaccine challenge: a randomised controlled trial. PLoS One. 2011 Mar 21;6(3):e14771. doi: 10.1371/journal.pone.0014771. PMID 21445287
- [Derived] Hurst R, Armah CN, Dainty JR, Hart DJ, Teucher B, Goldson AJ, Broadley MR, Motley AK, Fairweather-Tait SJ. Establishing optimal selenium status: results of a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2010 Apr;91(4):923-31. doi: 10.3945/ajcn.2009.28169. Epub 2010 Feb 24. PMID 20181815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ran from May until the following February in 2005, 2006, and 2007. Study completed in June 2008. 272 volunteers completed a screening questionnaire,182 volunteers had blood samples screened, total of 133 were recruited and 119 completed the study.
Groups:
- Placebo: Placebo
  Selenomethionine (supplement) and selenium enriched onions
Period: Overall Study
Arm/Group | Placebo | 50ug Selenium Enriched Yeast | 100ug Selenium Enriched Yeast | 200ug Selenium Enriched Yeast | Control Onion | Enriched Onion
Started | 21 | 26 | 24 | 23 | 20 | 19
Completed | 20 | 20 | 21 | 23 | 17 | 18
Not Completed | 1 | 6 | 3 | 0 | 3 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 50ug Selenium Enriched Yeast | 100ug Selenium Enriched Yeast | 200ug Selenium Enriched Yeast | Control Onion | Enriched Onion | Total
Number analyzed (Participants) | 20 | 20 | 21 | 23 | 17 | 18 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 21 | 23 | 17 | 18 | 119
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (3.9) | 56.5 (4.6) | 58.4 (3.9) | 56.1 (3.9) | 58.2 (5.1) | 57.7 (4.2) | 57.12 (1.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 11 | 11 | 6 | 6 | 54
  Male | 10 | 10 | 10 | 12 | 11 | 12 | 65
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 21 | 23 | 17 | 18 | 119
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25 (2.7) | 26.1 (3) | 26.3 (3.9) | 25.9 (3.8) | 26.6 (4.1) | 26.1 (2.4) | 26 (0.54)

OUTCOME MEASURES:

1. Primary Outcome: Cellular and Humoral Immune Response
Description: Total glutathione peroxidase 1 activity in platelets after supplementation
Time Frame: 12 weeks
Population: Data from 117 subjects because of incomplete time-course experiment for one subject and baseline plasma selenium concentration for one subject
Measure: Mean (Standard Deviation); unit: umol/min
Arm/Group | Placebo | 50ug Selenium Enriched Yeast | 100ug Selenium Enriched Yeast | 200ug Selenium Enriched Yeast | Control Onion | Enriched Onion
Number analyzed (Participants) | 20 | 18 | 21 | 23 | 17 | 18
umol/min | 0.29 (0.07) | 0.34 (0.16) | 0.34 (0.15) | 0.29 (0.09) | 0.35 (0.15) | 0.35 (0.13)
Statistical Analysis 1: Comparison: Placebo vs 50ug Selenium Enriched Yeast vs 100ug Selenium Enriched Yeast vs 200ug Selenium Enriched Yeast vs Control Onion vs Enriched Onion; Test type: Other; p < 0.05, ANOVA

2. Secondary Outcome: Selenium Status
Description: Plasma selenium concentration after supplementation
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | 50ug Selenium Enriched Yeast | 100ug Selenium Enriched Yeast | 200ug Selenium Enriched Yeast | Control Onion | Enriched Onion
Number analyzed (Participants) | 20 | 18 | 21 | 23 | 17 | 18
ng/mL | 93.7 (16.5) | 118.3 (13.1) | 152.0 (24.3) | 177.4 (26.3) | 94.2 (15.0) | 106.0 (11.9)
Statistical Analysis 1: Comparison: Placebo vs 50ug Selenium Enriched Yeast vs 100ug Selenium Enriched Yeast vs 200ug Selenium Enriched Yeast vs Control Onion vs Enriched Onion; Test type: Other; p = 0.05, Mixed Models Analysis

3. Secondary Outcome: Selenoproteins and Se-biomarkers
Description: Plasma selenoprotein P after the supllementation
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | 50ug Selenium Enriched Yeast | 100ug Selenium Enriched Yeast | 200ug Selenium Enriched Yeast | Control Onion | Enriched Onion
Number analyzed (Participants) | 20 | 18 | 21 | 23 | 17 | 18
ug/mL | 4.96 (0.86) | 6.17 (0.85) | 6.73 (1.01) | 6.59 (0.64) | 4.80 (1.03) | 5.72 (0.75)
Statistical Analysis 1: Comparison: Placebo vs 50ug Selenium Enriched Yeast vs 100ug Selenium Enriched Yeast vs 200ug Selenium Enriched Yeast vs Control Onion vs Enriched Onion; Test type: Other; p = 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | 50ug Selenium Enriched Yeast | 100ug Selenium Enriched Yeast | 200ug Selenium Enriched Yeast | Control Onion | Enriched Onion
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/26 | 0/24 | 0/23 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/26 | 0/24 | 0/23 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 1/26 | 1/24 | 0/23 | 2/20 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | 50ug Selenium Enriched Yeast (N=26) | 100ug Selenium Enriched Yeast (N=24) | 200ug Selenium Enriched Yeast (N=23) | Control Onion (N=20) | Enriched Onion (N=19)
cold symptoms (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No